CLINICAL TRIAL: NCT03245242
Title: Multicenter Pilot and Exploration Study of Enhanced Recovery After Surgery (ERAS) in Patients Undergoing Urologic Reconstructive Surgery
Brief Title: Pediatric Urology Recovery After Surgery Endeavor (PURSUE)
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201703081
Record Dates: First submitted 2017-07-28; First posted 2017-08-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Urologic Surgical Procedures; Urinary Bladder, Neurogenic; Urinary Bladder Diseases
Keywords: enhanced recovery after surgery; urologic reconstruction; pediatric urology; bladder augmentation; Mitrofanoff; Malone antegrade continence enema channel; appendicovesicostomy; ileovesicostomy; appendicocecostomy
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Bladder Diseases | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enhanced Recovery After Surgery: Prospectively enrolled group to receive standardized care under a set ERAS protocol/pathway.
  Interventions: Other: Enhanced Recovery after Surgery
- Historical usual surgical care: Recent historical patients (5 years prior to start of ERAS) that will be propensity-matched to ERAS patients to be used as controls for comparison of outcomes.
  Interventions: Other: Historical usual surgical care

INTERVENTIONS:
Other: Enhanced Recovery after Surgery — Enhanced Recovery After Surgery (ERAS) protocol is a multi-disciplinary program that aims to standardize care processes around the pre-, intra-, and post-operative care setting. This group will prospectively receive care under a pre-defined protocol.
  Groups: Enhanced Recovery After Surgery
Other: Historical usual surgical care — Recent historical controls will have received care under "usual care" that existed prior to implementation of an enhanced recovery protocol.
  Groups: Historical usual surgical care

SUMMARY:
The purpose of this research study is to evaluate an Enhanced Recovery After Surgery (ERAS) protocol in children and young adults undergoing urologic reconstructive surgery. The investigators plan to collect data on speed of recovery (how quickly pain improves, length of time in the hospital, and the need for additional pain control) on patients who receive care under the ERAS protocol and compare it to historical controls.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate Enhanced Recovery After Surgery (ERAS) in the pediatric setting for participants undergoing intraabdominal urologic reconstruction procedures. ERAS practices are being implemented in the department independent of research and this project will allow the investigators to review these practices.

Providers, participants, and family members will complete pre- and post- surgery questionnaires. These questionnaires are geared to collect demographic information about the participant and how the surgery affects their life situation. The providers will answer questions regarding their experience with ERAS.

Evidence-based ERAS principles and procedures are compulsory components of this project. These will be documented in the medical record and are considered standard of care practice as part of perioperative patient care.

Data collected from the medical record for each participant will aid in evaluating if adherence to the ERAS protocol is achieved.

ELIGIBILITY:
Inclusion criteria:

* Age greater than or equal to 4 or <26 years at time of surgery
* Undergoing urologic reconstructive surgery that includes primary bowel anastomosis (i.e., creation of continent ileovesicostomy [Monti], sigmoid Monti channel, enterocystoplasty)
* Undergoing urologic reconstructive surgery that includes possible bowel anastomosis (planned creation of continent appendicovesicostomy [Mitrofanoff] with inability to use appendix at time of surgery and creation of alternative channel requiring primary bowel anastomosis)

Exclusion criteria:

• Clinically constipated (defined as Bristol 1 or 2 stools more than once per week, bowel movement interval > every other day [e.g. only has bowel movement every 3 days, or palpable stool in > 50% of colon on physical preoperative exam)

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: There are 2 populations:
  1. ERAS patients: a. ages 4-17 and, b. transitional young adult 18-25
  2. Historical patients: a. ages 4-17 and, b. transitional young adult 18-25
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to ERAS protocol | 3 years
  Adherence to ERAS protocol items with # of items achieved (out of 20)

SECONDARY OUTCOMES:
Length of stay | 3 years
  Median primary inpatient hospital stay associated with surgery episode (# midnight)
Re-admissions within 30 days | 30 days
  Median number of re-admissions to any hospital within 30 days of surgery episode per patient
Re-operations within 90 days | 90 days
  Median number of unplanned re-operations within 90 days of surgery episode per patient
Number of visits to the emergency room within 90 day period | 90 days
  Median number of visits to any emergency room within 90 days of surgery episode per patient
Number of 30-day complications | 3 years
  Median number of 30-day complications by Clavien-Dindo classification per patient
Number of 90-day complications | 3 years
  Median number of 90-day complications by Clavien-Dindo classification per patient
Number of long-term complications within 1 year | 1 year
  Median number of long-term complications per patient
Daily IV morphine equivalents | 3 days after surgery
  Mean daily IV morphine equivalents (mg/kg) usage during first 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Coplen, M.D., Principal Investigator — Washington University School of Medicine
Locations (7):
- United States (7):
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Hospital of Richmond at Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore RP, Burjek NE, Brockel MA, Strine AC, Acks A, Boxley PJ, Chidambaran V, Vricella GJ, Chu DI, Sankaran-Raval M, Zee RS, Cladis FP, Chaudhry R, O'Reilly-Shah VN, Ahn JJ, Rove KO; PURSUE Study Group. Evaluating the role for regional analgesia in children with spina bifida: a retrospective observational study comparing the efficacy of regional versus systemic analgesia protocols following major urological surgery. Reg Anesth Pain Med. 2023 Jan;48(1):29-36. doi: 10.1136/rapm-2022-103823. Epub 2022 Sep 27. PMID 36167478
- [Derived] Rove KO, Strine AC, Wilcox DT, Vricella GJ, Welch TP, VanderBrink B, Chu DI, Chaudhry R, Zee RS, Brockel MA; PURSUE Study group. Design and development of the Pediatric Urology Recovery After Surgery Endeavor (PURSUE) multicentre pilot and exploratory study. BMJ Open. 2020 Nov 23;10(11):e039035. doi: 10.1136/bmjopen-2020-039035. PMID 33234633